CLINICAL TRIAL: NCT03891017
Title: Qualitative & Quantitative Comparison of Hydrostatic vs Vacuum Casting Methods in Trans-Tibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Heather Appling, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5180404
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hydrostatic Vacuum Casting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vacuum casting (Experimental): Vacuum casting will be performed using the Ottobock vacuum casting system. For our vacuum casting procedures, we will be following the protocols outlined in the Harmony Fabrication Quick Guide
  Interventions: Other: vacuum casting
- hydrostatic casting (Active Comparator): For the aqua casting system, we will be using an in-house manufactured device. This device will be created following guidelines from the PCAST Technical Manual
  Interventions: Other: hydrostatic casting

INTERVENTIONS:
Other: vacuum casting — Participants will be cast using vacuum casting (Ottobock Harmony) method. The method of casting will be randomized via RNG. Participants will be fitted with both sockets and dynamic alignment procedures will be performed. This 15-minute fitting and alignment period will address any extreme gait deviations and initial socket discomforts. After fitting, the participant will then be given a 15-minute adjustment period to wear the device. We will then begin the assessment phase, beginning with the timed Get-Up and Go test and followed by the 6-Minute Walk test. Each patient will perform 3 rounds of each test and patient order will be determined at random. The participants will be given a 10 min break between each series of tests. At the end, a questionnaire will be given.
  Arms: vacuum casting
Other: hydrostatic casting — Participants will be cast using aqua casting method. The method of casting will be randomized via RNG. Participants will be fitted with both sockets and dynamic alignment procedures will be performed. This 15-minute fitting and alignment period will address any extreme gait deviations and initial socket discomforts. After fitting, the participant will then be given a 15-minute adjustment period to wear the device. We will then begin the assessment phase, beginning with the timed Get-Up and Go test and followed by the 6-Minute Walk test. Each patient will perform 3 rounds of each test and patient order will be determined at random. The participants will be given a 10 min break between each series of tests. At the end, a questionnaire will be given.
  Arms: hydrostatic casting

SUMMARY:
The purpose of this graduate research study is to compare hydrostatic and vacuum casting techniques using patient mobility indicators, volume displacement, comfort, and overall satisfaction outcomes in trans-tibial amputees.

DETAILED DESCRIPTION:
Visit 1

* Informed Consent
* Subject will be casted using both the hydrostatic and vacuum system techniques

Visit 2 (7-10 days after Visit 1)

* One of two sockets will be randomly assigned and fitted/aligned by investigators
* Subject will be asked to perform a Timed Up and Go Test followed by a Six-Minute Walk Test
* Subject will fill out a comfort questionnaire for the prosthesis worn

Visit 3 (7 to 10 days after Visit 2)

• Subject will be asked to do the same testing as you performed in Visit 2

ELIGIBILITY:
Inclusion criteria :

* 18 years of age or older
* Trans-tibial amputation, unilateral
* Able to walk for a six-minute minimum w/o a break
* Amputation history of at least 6 months

Exclusion criteria:

* Syme amputation
* Physical disability or injury affecting a natural gait pattern
* Ulcers or blisters on the residual limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Six-Minute Walk Test | between 7-10- days after study enrollment
  Participants will walk in a 100-ft hallway on a flat, hard surface in a period of 6 minutes.

SECONDARY OUTCOMES:
Volume Calculation | between 7-10- days after study enrollment
  The Ohio Willow Wood Omega Tracer 3-dimensional image capture device and associated Omega shape capture software will be used to determine the volumes of each socket type, comparing the vacuum and aqua casting volume metrics. The scanning variables of width, depth, and length will determine the total displacement of each socket type. It has been determined that laser scanning is a valid and reliable method for accurately measuring volume fluctuations between casting methods.
Volume Calculation | between 14-20 days after study enrollment
  The Ohio Willow Wood Omega Tracer 3-dimensional image capture device and associated Omega shape capture software will be used to determine the volumes of each socket type, comparing the vacuum and aqua casting volume metrics. The scanning variables of width, depth, and length will determine the total displacement of each socket type. It has been determined that laser scanning is a valid and reliable method for accurately measuring volume fluctuations between casting methods.
Six-Minute Walk Test | between 14-20 days after study enrollment
  Participants will walk in a 100-ft hallway on a flat, hard surface in a period of 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Appling, MSOP, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No